CLINICAL TRIAL: NCT06356090
Title: Supportive Parenting for Anxious Childhood Emotions (SPACE): an Innovative Parent-based Treatment for Children With Obsessive-compulsive Disorder
Brief Title: SPACE: a Parent-based Treatment for Pediatric OCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chaim Huijser (Other)
Collaborators: Levvel (Unknown)
Responsible Party: Sponsor-Investigator, Chaim Huijser, Principal Investigator, Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023.0322 - NL84369.018.23
Record Dates: First submitted 2024-02-02; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Obsessive-Compulsive Disorder; Obsessive-Compulsive Disorder in Children; Obsessive-Compulsive Disorder in Adolescence; Anxiety Disorders and Symptoms
Keywords: SPACE; Family Accommodation; OCD; Anxiety; Children & adolescents; Parent-only treatment
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Single case experimental design (SCED) with multiple baselines
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPACE treatment with random baselines (Experimental): Participants are randomly allocated to one of three baseline periods (4 weeks, 6 weeks or 8 weeks). Only the parents of the participating families receive the SPACE treatment (12 sessions across 12 weeks). After the SPACE treatment, there is a follow-up period of 6 month after baseline.
  Interventions: Behavioral: Supportive Parenting for Anxious Childhood Emotions (SPACE)

INTERVENTIONS:
Behavioral: Supportive Parenting for Anxious Childhood Emotions (SPACE) — SPACE is a parent-based treatment (parent-stand-alone treatment) for parents of youth with anxiety symptoms or OCD. The manualized treatment protocol contains 12 sessions, in which parents are taught to reduce family accommodation (FA) and to increase supportive responses to their child.

SUMMARY:
This study will investigate the parent-based treatment SPACE: Supportive Parenting for Anxious Childhood Emotions. The aim of this study is to investigate whether SPACE is effective in reducing family accommodation (FA) and OCD symptoms in children with a complex obsessive-compulsive disorder (OCD), that did not or cannot benefit from first line treatment.

DETAILED DESCRIPTION:
Background:

Pediatric obsessive-compulsive disorder (OCD) is a severely impairing disorder where children experience anxiety or distress-provoking intrusive thoughts (obsessions) and/or engage in time-consuming ritualistic behaviours (compulsions). Approximately 40% of youth with OCD do not benefit from first-line treatment such as cognitive behavioral therapy (CBT) and pharmacotherapy. Family accommodation (FA) is highly prevalent in families of children affected by OCD. FA encompasses all behaviors of parents, siblings and other caregivers aimed to alleviate distress in the affected child. High levels of FA are associated with greater symptom severity, poorer functioning and inferior treatment outcomes in children and adolescents. However, FA is an under-addressed aspect in the treatment of children and adolescents. SPACE is a parent-based treatment where parents are taught to reduce FA and increase supportive responses towards the child, aiming to improve the child's OCD. An unique advantage of the program is that SPACE can be applied without cooperation of the child.

Objective:

The objectives of the present study are:

* to investigate whether SPACE is effective in reducing FA and OCD symptoms in children with complex OCD
* to explore mechanisms of change (in OCD symptoms) for the effectiveness of the SPACE treatment.

Method:

In this study, the investigators aim to include 25 Dutch children with OCD, their parent(s)/ caregiver(s) and their teacher.

To be eligible to participate in this study, subject must meet the following criteria: a) child (age 7-18 years) meets DSM-5 criteria for OCD (as primary classification) and meets the clinical cut-off score of 16 or higher for OCD on the Child Yale-Brown Obsessive Compulsive Scale (CY-BOCS) at baseline; b) previous psychosocial treatment for OCD was insufficient, child aborted treatment or was unable/ not motivated to receive treatment due to high level of anxiety/ OCD); c) Parents show high levels of FA at time of baseline on the Family Accommodation Scale Anxiety (FASA).

Medication use is allowed, provided that the medication regime had been stable for 4 weeks prior to participation and remains unchanged during participation.

Psychiatric comorbidity is allowed; however, a subject meeting any of the following criteria will be excluded for participation in this study: a) need for inpatient treatment; b) acute suicidality; c) psychotic symptoms d) no participating parents e) parents have insufficient mastery of the Dutch language f) parent or child has an estimated IQ below 75.

Design:

The current study will use a single-case experimental design (SCED) with multiple baselines. The course of the study will consist of a baseline phase, treatment phase and follow-up phase. Participating parents and their child will be randomized by computer to one of three baseline phase durations (4, 6 or 8 weeks). During the treatment phase, parents follow SPACE, which includes 12 treatment sessions provided by a trained and supervised professional. Throughout the different phases, there will be weekly measurements on FA and OCD symptoms, filled in by parents and children using a smartphone app. Semi-structured interviews will be conducted and questionnaires will be filled out by parents and children at T0 (baseline), T1 (start treatment), T2 (after 4 treatment sessions), T3 (after 8 treatment sessions), T4 (post treatment) and T5 (follow-up) and by teachers at T0, T4 and T5.

Analysis: For primary and secondary study outcomes visual data inspections will be performed to check for changes over time and between different phases of the SCED. A Reliable Change Index (RCI) will be calculated for changes in OCD symptoms and FA between pre- and post treatment assessments. Multilevel modeling will be used to test within-person changes over time. Meta-analysis will be performed over all included participants to test effects on group level. To explore mechanisms of change, cross-lagged correlations will be calculated to explore associations between two variables over time. Descriptive analysis will be used to determine predictors of treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* The child ages between 7 - 18 years old
* The child meets the DSM-5 criteria for OCD (as primary classification)
* The child did not benefit from psychological treatment for OCD (either followed 8 to 12 sessions of CBT or other psychotherapy), aborted treatment early or was unable/not motivated to receive treatment due to high levels of anxiety/OCD)
* At time of baseline still meets the clinical cut-off of 16 or higher for OCD on the Child Yale-Brown Obsessive Compulsive Scale [CY-BOCS].
* Psychiatric comorbidity is allowed, provided that OCD is the primary treatment target
* Parents report high levels of Family Accommodation (FA) at time of baseline (meeting the cut-off of 10 or higher on the Family Accommodation Scale Anxiety [FASA])
* Medication use is allowed. Selective serotonin reuptake inhibitors (SSRI) use (for OCD symptoms) is allowed as well, provided that the medication regime has been stable 4 weeks prior to participation and remains unchanged during participation.

Exclusion Criteria:

* The child needs inpatient treatment
* Acute suicidality
* Psychotic symptoms
* No participating parents
* Parents have insufficient mastery of the Dutch language
* Parents or child have an estimated IQ below 75

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
(Change in) OCD severity | Assessed at Timepoint 0 (start baseline), Timepoint 1 (start treatment: 4, 6 or 8 weeks after Timepoint 0), Timepoint 2 (± 4 weeks after T1), Timepoint 3 (± 8 weeks after Timepoint 1), Timepoint 4 (± 12 weeks after T1) & Timepoint 5 (6 months after T0)
  Measured using the Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS, a clinician rated semi-structured interview based on a combined parent and child-report). The CY-BOCS contains a severity scale and a symptom checklist. The symptom checklist assesses the current and past potential obsessive and compulsive experiences (indicated with 'yes' or 'no'). The severity scale consist of 5 items on obsession severity and 5 items on compulsion severity, rated on a Likert scale from 0 to 4. Higher scores represent more severity. The CY-BOCS Total Score is the sum of the obsession severity and compulsion severity items (range 0-40, with higher scores representing greater severity).
(Change in) family accommodation (parent report) | Assessed at Timepoint 0 (start baseline), Timepoint 1 (start treatment: 4, 6 or 8 weeks after Timepoint 0), Timepoint 2 (± 4 weeks after T1), Timepoint 3 (± 8 weeks after T1), Timepoint 4 (± 12 weeks after T1) & Timepoint 5 (6 months after T0)
  Measured using the Family Accommodation Scale Anxiety (FASA, parent version). Items are rated on a Likert scale from 0 to 4, with higher scores representing more family accommodation.
(Change in) Family accommodation (child report) | Assessed at Timepoint 0 (start baseline), Timepoint 1 (start treatment: 4, 6 or 8 weeks after Timepoint 0), Timepoint 2 (± 4 weeks after T1), Timepoint 3 (± 8 weeks after T1), Timepoint 4 (± 12 weeks after T1) & Timepoint 5 (6 months after T0)
  Measured using the Family Accommodation Scale Anxiety - Child Rated (FASA-CR, child version). Items are rated on a Likert scale from 0 to 4, with higher scores representing more family accommodation.
Daily (change in) OCD symptoms | 6 months - Assessed 3 times a week during 6 months
  Measured using two self-developed visual slider scales (rated on a 0-10 scale) in a mobile app (parents and child-report). Higher scores indicate more perceived OCD symptoms and more time spent on OCD symptoms.
Daily (change in) family accommodation | 6 months - Assessed 3 times a week during 6 months
  Measured using two self-developed visual slider scales (rated on a 0-10 scale) in a mobile app (parents and child-report). Higher scores indicate more perceived FA and more time spent on FA.

SECONDARY OUTCOMES:
Symptoms of child anxiety | Assessed at Timepoint 0 (start baseline), Timepoint 1 (start treatment: 4, 6 or 8 weeks after Timepoint0), Timepoint 4 (± 12 weeks after T1) & Timepoint 5 (6 months after T0)
  Measured using the Screen for Childhood Anxiety Related Emotional Disorder- NL (SCARED-NL, child-report). Items are rated on a scale from 0-2. The total score on the SCARED ranges form 0-138. Higher scores indicate more severe anxiety.
Symptoms of child depression | Assessed at Timepoint 0 (start baseline), Timepoint 1 (start treatment: 4, 6 or 8 weeks after Timepoint0), Timepoint 4 (± 12 weeks after T1) & Timepoint 5 (6 months after T0)
  Measured using the Children Depression Inventory-2 (CDI-2, child-report). Items are rated on a scale from 0-2. The total score ranges from 0-56. Higher scores indicate more severe depressive symptoms.
Symptoms of autism | Assessed at Timepoint 0 (start baseline)
  Measured using the Social Responsiveness Scale (SRS-2, parent-report). Items are rated on a scale from 0-3. The total score ranges from 0-195. Higher scores indicate greater autism symptom severity.
Quality of life (parent-report) | Assessed at Timepoint 0 (start baseline), Timepoint 4 (± 12 weeks after Timepoint 1) & Timepoint 5 (6 months after Timepoint 0)
  Measured using the EuroQol 5D (EQ-5D, adult version), consisting the EQ-5D Index and the EQ Visual Analog Scale (EQ VAS). There a 5 predefined dimensions: Mobility, Self-care, Usual activities, Pain/ Discomfort and Anxiety/ Depression. Items are rated on a 3 level scale. The EQ VAS score is rated on a visual analogue scale ranging from 0 ('the worst health you can imagine') to 100 ('the best health you can imagine').
Quality of life (child-report) | Assessed at Timepoint 0 (start baseline), Timepoint 4 (± 12 weeks after Timepoint 1) & Timepoint 5 (6 months after Timepoint 0)
  Measured using the EuroQol 5D-Youth (EQ-5D-Y, child-version), consisting the EQ-5D-Y descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive symptom comprises 5 dimensions: Mobility, Looking after myself, Doing usual activities, Having pain or discomfort and Feeling worried, sad or unhappy. Each dimension can be rated on 3 levels: no problems, some problems and a lot of problems. The EQ VAS records the respondent's self-rated health on a visual analogue scale ranging from 0 ('The best health you van imagine') to100 ('The worst health you can imagine').
Clinical impression of outcome | 3 months - Assessed weekly after each treatment session
  Measured using the Clinical Global Impression scale (CGI, clinician-report). The CGI comprises two one-item measures evaluating: 1) the severity of psychopathology rated on a scale from 0 (no symptoms) to 7 (extremely severe symptoms) and 2) change from the initiation of treatment on a similar scale from 0 (very much improved since initiation of treatment) to 7 (very much worse since the initiation of treatment).
Treatment progress | During the intervention of 3 month, assessed before the start of each treatment session
  Treatment progress is measured using the Outcome Rating Scale (ORS, parent-report). The ORS comprises 4 short questions rated on a visual analog scale from 0 to 10. Higher scores indicate greater mental health during treatment.
Session experience | During the intervention of 3 month, assessed after each treatment session
  Person's overall therapy experience is measured using the Session Rating Scale (SRS, parent-report). The SRS comprises 4 short questions on a visual analog scale from 0 to10. Higher scores indicate greater satisfaction with the therapeutic alliance.
Treatment adherence | During the intervention of 3 months, rated after each treatment session
  Checklist for therapist, with checkboxes indicating adherence to treatment components.

OTHER OUTCOMES:
Demographic variables | Assessed at Timepoint 0 (start baseline)
  Such as gender, age of the child, cultural background, family functioning, educational level and life events (parent-report).
Psychiatric DSM-5 diagnosis of the child | Assessed at Timepoint 0 (start baseline), Timepoint 4 (± 12 weeks after Timepoint 1) & Timepoint 5 (6 months after Timepoint 0)
  Measured using the Structured Clinical Interview for DSM-5 Childhood Disorders (SCID-5 junior) (parent and child interview, clinician-rated). Clinicians rate the presence or absence of DSM-5 diagnosis.
Parenting burden | Assessed at Timepoint 0 (start baseline), Timepoint 4 (± 12 weeks after Timepoint 1) & Timepoint 5 (6 months after Timepoint 0)
  Measured using the Stress of Parenting Questionnaire (OBVL, parent-report). Items are rated on a scale from 1 to 4. The total score ranges from 34 to 136, with higher scores indicating greater parental burden.
Psychopathology and adaptive functioning of parents | Assessed at Timepoint 0 (start baseline), Timepoint 4 (± 12 weeks after Timepoint 1) & Timepoint 5 (6 months after Timepoint 0)
  Measured using the Achenbach System of Empirically Based Assessment - Adult Self Report (ASEBA -ASR, parent-report). Items are rated on a scale from 0 ('not true') to 2 ('very true or often true'). The Total Problem score on the ASR, based on 120 problem items, ranges from 0 to 240. Higher scores indicate more problems related to adult psychopathology.
Child Behavior Checklist (CBCL, parent-report) | Assessed at Timepoint 0 (start baseline), Timepoint 4 (± 12 weeks after Timepoint 1) & Timepoint 5 (6 months after Timepoint 0)
  The Child Behavior Checklist, part of the Achenbach System of Empirically Based Assessment (ASEBA - CBCL), is a parent reported questionnaire that consists 118 items that seek to assess behavioral and emotional problems in children from 6 to 18 years old. Items are rated on a 3-point scale: 0 = 'not true', 1 = 'somewhat or sometimes true' and 2 = 'very true or often true'. It comprises three scales: (1) Internalizing problems; (2) Externalizing problems; (3) Total problem score. Higher scores indicate more emotional- and behavioral problems reported by the parent. On all scales, T-Score = 60 or more indicates a clinical level of the child's emotional and behavioral problems.
Youth Self-report (YSR) (child-report) | Assessed at Timepoint 0 (start baseline), Timepoint 4 (± 12 weeks after T1) & Timepoint 5 (6 months after T0)
  The Youth Self-report, part of the Achenbach System of Empirically Based Assessment (ASEBA - YSR), is a child reported questionnaire that consists 112 items that seek to assess behavioral and emotional problems in children from 11 to 18 years old. Items are rated on a 3-point scale: 0 = 'not true', 1 = 'somewhat or sometimes true' and 2 = 'very true or often true'. Higher scores indicate more emotional- and behavioral problems reported by the child. It comprises three scales: (1) Internalizing problems; (2) Externalizing problems; (3) Total problem score. On all scales, T-Score = 60 or more indicates a clinical level of the child's emotional and behavioral problems.
Teacher Report Form Emotional- and behavioral problems of the child (teacher- report) | Assessed at Timepoint 0 (start baseline), Timepoint 4 (± 12 weeks after Timepoint 1) & Timepoint 5 (6 months after Timepoint 0)
  Measured using the Achenbach System of Empirically Based Assessment - Teacher Report Form (ASEBA - TRF, teacher-report). Items are rated on a 3-point scale: 0 = 'not true', 1 = 'somewhat or sometimes true' and 2 = 'very true or often true'. Higher scores indicate more emotional- and behavioral problems reported by the teacher. It comprises three scales: (1) Internalizing problems; (2) Externalizing problems; (3) Total problem score. Higher scores indicate more emotional- and behavioral problems reported by the parent. On all scales, T-Score = 60 or more indicates a clinical level of the child's emotional and behavioral problems.
Treatment satisfaction | Timepoint 4 (± 12 weeks after Timepoint 1)
  Measured using a self-developed questionnaire on treatment preferences and satisfaction (11 questions, parent-report). Items are rated on a scale from 1 to 5, with higher scores indicating greater treatment satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: C. Huijser, Dr., Principal Investigator — Amsterdam UMC / Levvel
Locations (1):
- Amsterdam UMC / Levvel (Academic centre for child & adolescent psychiatry), Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data will not be openly and publically available, since the data is sensitive. Qualified researchers can request access to anonymized individual participant data for research purposes such as meta-analyses, and questionnaire validation studies. An encrypted, merged and prepared dataset can be made available for re-use in line with the FAIR (Findable, Accessible, Interoperable, and Reusable) data principles. The Principle Investigator is responsible for the data and can be contacted for requests after completion and publication of the present study. Participant will be asked informed consent for re-use and sharing of the anonymous individual participant data. An agreement will be drawn up, when data sharing is requested.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After completion and publication of the present study, data sharing can be requested.
Access Criteria: Requests for data sharing will be assessed by the Principal Investigator.

REFERENCES:
- [Background] Lebowitz ER, Marin C, Martino A, Shimshoni Y, Silverman WK. Parent-Based Treatment as Efficacious as Cognitive-Behavioral Therapy for Childhood Anxiety: A Randomized Noninferiority Study of Supportive Parenting for Anxious Childhood Emotions. J Am Acad Child Adolesc Psychiatry. 2020 Mar;59(3):362-372. doi: 10.1016/j.jaac.2019.02.014. Epub 2019 Mar 7. PMID 30851397
- [Background] Maric M, Werff V. Single-Case Experimental Designs in Clinical Intervention Research. Small Sample Size Solutions. 2020;102-111.